CLINICAL TRIAL: NCT03356197
Title: Epidemiology of Conjunctivitis in the Emergency Department of a Reference Ophthalmological Hospital in Goiânia
Brief Title: Epidemiology of Conjunctivitis in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: Conjuntivite ARVO 2018
Record Dates: First submitted 2017-11-19; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Acute Conjunctivitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiology of Conjunctivitis in the Emergency Department of a Reference Ophthalmological Hospital in Goiânia.

DETAILED DESCRIPTION:
The purpose of this study was to determine the epidemiology of ocular emergencies in a Reference Ophthalmological Hospital in Goiânia, with emphasis on acute infectious conjunctivitis, morbidity with a higher incidence in this Service. It aims to delineate the main etiologies found among infectious conjunctivitis and to compare them with those found in several other reference services in Ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

* All those patients who were submitted to a initial care performed by the First Year Resident (R1) of the Hospital and who were admitted during the period described.

Exclusion Criteria:

* The patients who were admitted in the Emergency Department outside this period
* The patients who were not attended by a First Year Resident (R1)
* The patients who did not have all the data filled in the medical record
* The patients who needed to return, being attended in the hospital more than once.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were submitted to a initial care in the Emergency Department performed by the Ophthalmology First Year Resident (R1) .
Sampling Method: Non-Probability Sample
Enrollment: 783 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the main etiologies of acute infectious conjunctivitis in the Emergency Department of a Reference Hospital in Goiânia. | 126 days
  Through clinical diagnosis in the Emergency Department

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil